CLINICAL TRIAL: NCT04331743
Title: A Single-arm, Open-label, Single-center Phase Ib Study to Evaluate the Safety and Efficacy of Liposome-entrapped Mitoxantrone Hydrochloride Injection (PLM60) in Advanced Hepatocellular Carcinoma (HCC)
Brief Title: A Study to Evaluate the Safety and Efficacy of PLM60 in Advanced HCC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLM60-HCC-201901/PRO
Record Dates: First submitted 2020-03-12; First posted 2020-04-02 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Advanced Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLM60 (Experimental): Three dose levels will be tested according to the "3 + 3" dose-escalation design.The dose-limiting toxicity (DLT) will be assessed from the first administration of PLM60 to the end of the first cycle (28 days).
  Interventions: Drug: Liposome-entrapped Mitoxantrone Hydrochloride Injection

INTERVENTIONS:
Drug: Liposome-entrapped Mitoxantrone Hydrochloride Injection — Intravenous infusion
  Other Names: PLM60

SUMMARY:
This is a dose escalation study based on 3+3 design with the aim to establish MTD and provide RP2D. PLM60 is to administered by multi-cycle intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from the patient；
* ECOG performance status of 0 or 1;
* Histologically/cytologically confirmed diagnosis of advanced HCC;
* Adequate washout period for previous anti-tumor therapy;
* Measurable disease according to RECIST v1.1;
* Life expectancy ≥ 12 weeks;
* Adequate organ function;
* Child-Pugh grade A or partial grade B; BCLC stage B or C;V

Exclusion Criteria:

* Prior treatment with Mitoxantrone or Liposome-entrapped Mitoxantrone, or other anthracyclines, with the total cumulative dose of > 360 mg/m2 ;
* Any drug-related adverse event derived from any previous anti-tumor treatment, excluding alopecia, Pigmentation, or other toxicity with little safety risk for subjects, that has not recovered to grade1 or less;
* Active central nervous system (CNS) metastases (brain or leptomeningeal metastases, etc.);
* Any history of other malignancy within 5 years;
* Untreated hepatitis infection;
* HIV positive;
* History of liver transplantation, severe cirrhosis, hepatic encephalopathy;
* Inadequate cardiac function;
* Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-06-05 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limited toxicity (DLT) | 1year
  To identify the dose-limited toxicity (DLT).
Maximum tolerated dose (MTD) | 1 year
  To identify the maximum tolerated dose (MTD).
Recommended Phase II Dose (RP2D) | 1 year
  To identify the Recommended Phase II Dose (RP2D)

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 2 years
  To preliminarily evaluate the AUC in patients with advanced HCC.
Peak Plasma Concentration (Cmax) | 2 years
  To preliminarily evaluate Cmax in patients with advanced HCC.
Time of peak plasma concentration (Tmax) | 2 years
  To preliminarily evaluate Tmax in patients with advanced HCC.
Median overall survival (OS) | 2 years
  To preliminarily evaluate ORR in patients with advanced HCC.
Median progression free survival (PFS) | 2 years
  To preliminarily evaluate PFS in patients with advanced HCC.
Overall response rate (ORR) | 2 years
  To preliminarily evaluate ORR in patients with advanced HCC.
Duration of Response (DoR) | 2 years
  To preliminarily evaluate DoR in patients with advanced HCC.

IPD SHARING:
Plan to Share IPD: Undecided